CLINICAL TRIAL: NCT01269593
Title: PET Imaging of Cancer Patients Using 124I-PUH71: A Pilot Study
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Samus Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-139
Record Dates: First submitted 2010-12-29; First posted 2011-01-04 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin's Lymphoma; Myeloma; Active Solid Malignancy
Keywords: PET Scan; 124I-PUH71; 10-139
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell

ARMS (1):
- PET Imaging Using 124 IPUH71 (Experimental): Patients will receive an injection of up to 11.0 mCi (range: 4.0-11.0 mCi) of 124I-PUH71, followed by serial PET scanning and blood draws, over a period of 3 days. Optional with a fourth day of PET scanning is to be pursued, in willing patients.
  Interventions: Drug: PET Imaging using 124 IPUH71

INTERVENTIONS:
Drug: PET Imaging using 124 IPUH71 — A dose of up to 11.0 mCi (range: 4.0-11.0 mCi) of 124I-PUH71 will be administered intravenously with the patient at rest. 124I-PUH71 scans will be performed at immediately and/or 3-4 hours, 20-24 hours, and 40-80 hours after injection of the radiotracer. Optionally, in willing patients scans will be performed 160-200 hours (~7-8 days) after injection of the radiotracer. At each time-point, a 45-60 minute axial body image is acquired. Images will be acquired on a state-of-the-art PET-CT scanner. A low-dose CT will be obtained immediately-prior to PET imaging, at each time-point. A 30-45 minute scanning timeperiod is typical for clinical PET studies.
  Other Names: Blood will be drawn at the multiple time points for pharmacokinetic & metabolite; analyses of 124I-PUH71. We anticipate these time points to be: approximately 10; minutes, 20 minutes, 30 minutes, 1-2 H, and 3-4 H, post-injection. Blood; samples will be obtained in the PET imaging suite.

SUMMARY:
The purpose of this study is to see how a new drug, named PUH71, accumulates in the different parts of the body & inside tumors and how long PUH71 lasts in the blood, when given to study participants in tiny amounts. The results of this study will help researchers (1) plan how they will use PUH71 as an experimental new drug (at much-higher doses) for the treatment of cancer, in clinical trials; and (2) know whether PUH71 might be used as a drug for detecting tumors with scanner machines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid malignancy, myeloproliferative neoplasm, myeloma, and/or lymphoma (histology confirmed by MSKCC Department of Pathology)
* Disease is measurable or evaluable as defined by RECIST (1.1 or original version) or other tumor response criteria from an MSKCC IRB-approved clinical research protocol.
* This does not apply to patients with myeloproliferative neoplasm. The presence of active myeloproliferative neoplasm will be determined by applicable disease specific diagnostic criteria and patient assessment by the patient's oncologist and trial investigators (eg, manifestations of active MPN such as splenomegaly, abnormal blood counts, etc).
* Age between 18-90
* Negative serum pregnancy test for females of childbearing age (11-55 years) and/or lack child-bearing potential
* No breast-feeding

Exclusion Criteria:

* Previous allergic reaction to contrast medium.
* Hypersensitivity to iodide products.
* Known hyperthyroidism

Hepatic:

* Bilirubin > 1.5 x institutional upper limit of normal (ULN)
* AST/ALT >2.5 x ULN
* Albumin < 2 g/dl
* GGT > 2.5 x ULN IF Alkaline phosphatase > 2.5 x ULN. Renal: Creatinine >1.5 x ULN or creatinine clearance < 60 mL/min.
* Positive serum pregnancy test for females
* Acute major illness (e.g., infection, unstable cardiovascular condition, etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To study the pharmacokinetics | 2 years
  of 124I-PUH71 in patients with solid malignancy, myeloproliferative neoplasm, myeloma, and/or lymphoma.

SECONDARY OUTCOMES:
To study the metabolism | 2 years
  of 124I-PUH71 in patients with solid malignancy, myeloproliferative neoplasm myeloma and/or lymphoma.
To study the biodistribution | 2 years
  of 124I-PUH71 in patients with solid malignancy, myeloproliferative neoplasm myeloma and/or lymphoma.
To study the radiation dosimetry | 2 years
  of 124I-PUH71 in patients with solid malignancy, myeloproliferative neoplasm myeloma and/or lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dunphy, DO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm